CLINICAL TRIAL: NCT03838198
Title: Developing an Adaptive Intervention for Suicidal Adolescents Following Inpatient Hospitalization: A Pilot SMART
Brief Title: An Adaptive Intervention for Adolescents at Risk for Suicide: A Pilot SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ewa Czyz, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HUM00129173; 1K23MH113776-01 (NIH)
Record Dates: First submitted 2019-02-06; First posted 2019-02-12 (Actual); Results first posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Suicide; Self Harm
Keywords: Adaptive Intervention; Sequential, Multiple Assignment, Randomized Trial (SMART); Adolescent; Motivational Interviewing; Suicide attempt; Safety planning; mobile technology
MeSH Terms: conditions — Suicide; Self-Injurious Behavior; Suicide, Attempted

STUDY DESIGN:
Intervention Model Description: This Sequential, Multiple Assignment, Randomized Trial (SMART) pilot of a Motivational Interview (MI)-enhanced safety planning intervention is designed to inform the development of a technology-augmented adaptive intervention for youth at risk for suicide. The MI-SafeCope intervention includes three components: (1) MI-enhanced safety plan delivered during hospitalization (encompassing individual and family meetings); (2) post-discharge booster call; and (3) post-discharge daily text message boosters. In this SMART pilot, adolescents will be randomized to either MI-enhanced safety plan alone or in combination with text boosters for two weeks after discharge (Phase 1 intervention). At the end of week 2, adolescents will be re-randomized to two additional weeks of either: continuation of Phase 1 intervention or continuation of Phase 1 intervention with the addition of post-discharge booster call. Thus, participants will receive one of four treatment sequences (Groups A-D).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Safety plan + booster text messages + booster call (Group A) (Other): Sequencing of MI-SafeCope intervention components (Phase 1 and Phase 2) resulting in Group A: Participants will receive the in-person MI-enhanced safety plan (individual meeting with the adolescent and a family meeting) during hospitalization -- focused on developing a personalized list of coping strategies and enhancing adolescents' motivation and self-efficacy to utilize these strategies-- which will be followed by 4 weeks of daily post-discharge booster text messages and a phone booster call.
  Interventions: Behavioral: MI-Enhanced Safety Plan at Hospitalization (1st Component); Behavioral: MI-Enhanced Text Boosters (2nd Component); Behavioral: MI-Enhanced Booster Call (3rd Component)
- Safety plan + booster text messages (Group B) (Other): Sequencing of MI-SafeCope intervention components (Phase 1 and Phase 2) resulting in Group B: Participants will receive the in-person MI-enhanced safety plan during hospitalization followed by 4 weeks of daily booster text messages post discharge.
  Interventions: Behavioral: MI-Enhanced Safety Plan at Hospitalization (1st Component); Behavioral: MI-Enhanced Text Boosters (2nd Component)
- Safety plan + booster call (Group C) (Other): Sequencing of MI-SafeCope intervention components (Phase 1 and Phase 2) resulting in Group C: Participants will receive the in-person MI-enhanced safety plan during hospitalization followed by a post-discharge booster call.
  Interventions: Behavioral: MI-Enhanced Safety Plan at Hospitalization (1st Component); Behavioral: MI-Enhanced Booster Call (3rd Component)
- Safety plan (Group D) (Other): Sequencing of MI-SafeCope intervention components (Phase 1 and Phase 2) resulting in Group D: Participants will receive the in-person MI-enhanced safety plan during hospitalization.
  Interventions: Behavioral: MI-Enhanced Safety Plan at Hospitalization (1st Component)

INTERVENTIONS:
Behavioral: MI-Enhanced Safety Plan at Hospitalization (1st Component) — The MI-enhanced safety plan intervention component is delivered during hospitalization and includes an individual and family meetings. The goal of the individual meeting with the adolescent is to develop an individualized safety plan for use during a suicidal crisis. This "best practices" approach of safety planning is augmented with Motivational Interviewing (MI) as a core strategy to explicitly elicit adolescents' motivation and commitment to behavior change (i.e. use safety plan; adaptive coping), address barriers or ambivalence, and strengthen self-efficacy. The focus of the family meeting, which is similarly guided by MI, is to prepare parents/guardians, with input from the adolescent, for how they may support the adolescent in implementing the individualized safety plan after discharge and on strengthening parents' commitment and self-efficacy.
Behavioral: MI-Enhanced Text Boosters (2nd Component) — For participants randomized to receive text boosters, booster text messages will be sent daily for 4 weeks. The messages will be tailored to encourage use of individualized coping strategies identified as part of safety planning at hospitalization and will include additional adaptive coping tools and resources. The text message content and tone will be consistent with principles of MI.
  Arms: Safety plan + booster text messages (Group B); Safety plan + booster text messages + booster call (Group A)
Behavioral: MI-Enhanced Booster Call (3rd Component) — The focus of the post-discharge booster phone call with adolescent and with parent, each conducted separately, will be to to further adjust the safety plan to better meet post-discharge needs, to further enhance adolescents' motivation and commitment to use coping strategies, and to further support adolescents' and parents' self-efficacy to manage suicidal crises.
  Arms: Safety plan + booster call (Group C); Safety plan + booster text messages + booster call (Group A)

SUMMARY:
To inform the development of a technology-augmented adaptive intervention for adolescents at risk for suicide, the goal of this study is to conduct a Sequential, Multiple Assignment, Randomized Trial (SMART) pilot of a Motivational Interview (MI)-enhanced safety planning intervention (MI-SafeCope). Findings from this study will provide the groundwork for the construction of a technology-augmented adaptive intervention that could lead to a reduction in suicidal behaviors and related events during the high-risk post-discharge period-an important suicide prevention target.

ELIGIBILITY:
Inclusion Criteria:

* Suicide attempt (previous month), and/or
* Suicidal ideation (previous week)

Exclusion Criteria:

* Severe cognitive impairment or altered mental status (psychosis, manic state)
* Transfer to medical unit or residential placement
* No availability of a legal guardian
* No cell phone with text messaging capability

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2020-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Czyz, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Czyz EK, King CA, Prouty D, Micol VJ, Walton M, Nahum-Shani I. Adaptive intervention for prevention of adolescent suicidal behavior after hospitalization: a pilot sequential multiple assignment randomized trial. J Child Psychol Psychiatry. 2021 Aug;62(8):1019-1031. doi: 10.1111/jcpp.13383. Epub 2021 Feb 15. PMID 33590475

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of a larger number of hospital admissions records reviewed, 94 persons were deemed "eligible" and were approached. 82 consented to participate in the trial, of whom, two participants were consented but excluded prior to randomization because they were discharged early.
Groups:
- Safety Plan + Booster Text Messages + Booster Call: Sequencing of MI-SafeCope intervention components (Phase 1 and Phase 2) resulting in Group A: Participants will receive the in-person MI-enhanced safety plan (individual meeting with the adolescent and a family meeting) during hospitalization -- focused on developing a personalized list of coping strategies and enhancing adolescents' motivation and self-efficacy to utilize these strategies -- which will be followed by 4 weeks of daily post-discharge booster text messages and in Period/Phase 2 a phone booster call.
- Safety Plan + Booster Text Messages: Sequencing of MI-SafeCope intervention components (Phase 1 and Phase 2) resulting in Group B: Participants will receive the in-person MI-enhanced safety plan during hospitalization followed by 4 weeks of daily booster text messages post discharge without booster phone call.
- Safety Plan + Booster Call: Sequencing of MI-SafeCope intervention components (Phase 1 and Phase 2) resulting in Group C: Participants will receive the in-person MI-enhanced safety plan during hospitalization followed by a post-discharge booster call.
- Safety Plan: Sequencing of MI-SafeCope intervention components (Phase 1 and Phase 2) resulting in Group D: Participants will receive the in-person MI-enhanced safety plan during hospitalization with neither follow-up text messages nor booster phone call.
Period: Phase 1: Safety Plan (SP) vs. SP w/Texts
Arm/Group | Safety Plan + Booster Text Messages + Booster Call | Safety Plan + Booster Text Messages | Safety Plan + Booster Call | Safety Plan
Started | 0 (Because it was a SMART trial, no participants were allocated to receive booster calls until Phase 2.) | 40 | 0 (Because it was a SMART trial, no participants were allocated to receive booster calls until Phase 2.) | 40
Completed | 0 | 40 | 0 | 40
Not Completed | 0 | 0 | 0 | 0
Period: Phase 2: Added Booster Call or Not
Arm/Group | Safety Plan + Booster Text Messages + Booster Call | Safety Plan + Booster Text Messages | Safety Plan + Booster Call | Safety Plan
Started (Started here means randomized in Phase 2 to either booster call or no booster call.) | 18 (These participants continued with Phase 1 intervention (Safety plan and text) with added booster call.) | 22 (These participants continued with Phase 1 intervention (Safety plan and text) with no added booster call.) | 18 (These participants continued with Phase 1 intervention (Safety plan only) with added booster call.) | 22 (These participants continued with Phase 1 intervention (Safety plan only) with no added booster call in Phase 2)
Completed | 18 (All 18 completed the safety plan; but only 14 had both parent and adolescent completing the call; 1 had parent only; 1 had adolescent only; 2 were unable to be reached.) | 0 | 17 (Of the 17 who completed the safety plan, only 15 had both parent and adolescent completing the call; 1 had parent only; 1 was unable to be reached.) | 0
Not Completed | 0 | 22 | 1 | 22
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — In this SMART trial design, this group was randomized to "no booster call. | 0 | 22 | 0 | 22
Period: 1 Month Follow up Period
Arm/Group | Safety Plan + Booster Text Messages + Booster Call | Safety Plan + Booster Text Messages | Safety Plan + Booster Call | Safety Plan
Started | 18 | 22 (All participants from Phase 1 and 2 were followed unless they withdrew.) | 17 | 22 (All participants from Phase 1 and 2 were followed unless they withdrew.)
Adolescent Surveys Completed | 16 | 22 | 16 | 22
Completed (Completed means parent survey completed) | 16 | 22 | 16 | 21
Not Completed | 2 | 0 | 1 | 1
Period: 3 Month Follow up Period
Arm/Group | Safety Plan + Booster Text Messages + Booster Call | Safety Plan + Booster Text Messages | Safety Plan + Booster Call | Safety Plan
Started (All participants (except the one who withdrew) were recontacted for 3 month follow up.) | 18 | 22 | 17 | 22
Adolescent Survey Completed | 16 | 21 | 15 | 21
Completed (Completed means parent survey completed) | 15 | 19 | 14 | 18
Not Completed | 3 | 3 | 3 | 4

BASELINE CHARACTERISTICS:
Population: Phase 1 assigned all 80 participants to safety plan(SP) or SP+text. Phase 2 added booster calls vs. no calls to Phase 1 interventions. Each participant of the 80 is fully included in the two groups shown here. For race, some participants self-described in >1 category, not as "More than 1 race". Thus the totals of participants' self-descriptions for race in each column exceed the actual 40 people shown in other baseline measures.
Groups:
- Phase 1 - Safety Plan: Participants who received the in-person MI-enhanced safety plan (individual meeting with the adolescent and a family meeting) during hospitalization -- focused on developing a personalized list of coping strategies and enhancing adolescents' motivation and self-efficacy to utilize these strategies
- Phase 1 - Safety Plan & Text Messages: Participants who received the in-person MI-enhanced safety plan during hospitalization followed by 4 weeks of daily booster text messages post discharge.
- Total: Total of all reporting groups
Arm/Group | Phase 1 - Safety Plan | Phase 1 - Safety Plan & Text Messages | Total
Number analyzed (Participants) | 41 | 42 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: This is the actual number of participants assigned to this group
  years
    number analyzed (Participants) | 40 | 40 | 80
    (all) | 15.08 (1.4) | 15.25 (1.32) | 15.16 (1.35)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: This is the actual number of participants assigned to this group
  Participants
    number analyzed (Participants) | 40 | 40 | 80
    Female | 27 | 27 | 54
    Male | 13 | 13 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: For race, some of the 40 participants assigned to each safety plan group self-described as more than one category, but not as "More than one race" . Thus the totals of participants' self-descriptions for race in each column total more than the overall number of baseline participants.
  Participants
    American Indian or Alaska Native | 3 | 1 | 4
    Asian | 2 | 2 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Black or African American | 3 | 2 | 5
    White | 32 | 35 | 67
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 1 | 1 | 2
Count of participants with at least one suicide attempt during their lifetime [Count of Participants; unit: Participants] — Population: This is the actual number of participants assigned to this group
  Participants
    number analyzed (Participants) | 40 | 40 | 80
    (all) | 21 | 19 | 40
Last-month suicide attempt [Count of Participants; unit: Participants] — Population: This is the actual number of participants assigned to this group
  Participants
    number analyzed (Participants) | 40 | 40 | 80
    (all) | 18 | 12 | 30
Multiple attempt history [Count of Participants; unit: Participants] — Population: This is the actual number of participants assigned to this group
  Participants
    number analyzed (Participants) | 40 | 40 | 80
    (all) | 14 | 14 | 28
Lifetime nonsuicidal self-injury [Count of Participants; unit: Participants] — Population: This is the actual number of participants assigned to this group
  Participants
    number analyzed (Participants) | 40 | 40 | 80
    (all) | 31 | 31 | 62
Suicidal ideation mean [Mean (Standard Deviation); unit: units on a scale] — Suicidal Ideation (Columbia-Suicide Severity Rating Scale (C-SSRS)) is scored on a range from 0 (no suicidal ideation) to 5 (suicidal ideation with plan and intent). Population: This is the actual number of participants assigned to this group
  units on a scale
    number analyzed (Participants) | 40 | 40 | 80
    (all) | 3.90 (.90) | 3.93 (0.92) | 3.91 (0.90)
Common Diagnoses [Count of Participants; unit: Participants] — Population: This is the actual number of participants assigned to this group
  Participants
    Depressive disorder: number analyzed (Participants) | 40 | 40 | 80
    Depressive disorder | 32 | 37 | 69
    Anxiety disorder: number analyzed (Participants) | 40 | 40 | 80
    Anxiety disorder | 20 | 23 | 43

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eligible Participants Recruited to the Study
Description: Eligible participants were candidates for participation based on medical record review who were approached for consent/assent.
  The percentage of eligible participants who consented to the study is presented below.
Time Frame: At time of study enrollment, measured following study consent/assent
Population: Eligible youth whether consent was provided or not
Measure: Number; unit: Percentage of eligible participants
Groups:
- All Eligible Youth: Potential participants prior to randomization
Arm/Group | All Eligible Youth
Number analyzed (Participants) | 94
Percentage of eligible participants | 87.2

2. Primary Outcome: Percentage of Randomized Participants Who Complete Intervention Components Will be Used to Assess Feasibility and Acceptability
Description: Outcome measure is showing percentage of randomized adolescent participants who complete intervention components to assess feasibility and acceptability
Time Frame: Following intervention, measured up to 1 month
Population: No texts and boosters were planned for the associated data fields
Measure: Number; unit: percent of participants
Arm/Group | Safety Plan + Booster Text Messages + Booster Call (Group A) | Safety Plan + Booster Text Messages (Group B) | Safety Plan + Booster Call (Group C) | Safety Plan (Group D)
Number analyzed (Participants) | 18 | 22 | 18 | 22
percent of participants
  Safety Plan (Phase 1) | 100 | 100 | 100 | 100
  Booster Texts: number analyzed (Participants) | 18 | 22 | 0 | 0
  Booster Texts | 100 | 100 |  |
  Booster Call (Phase 2): number analyzed (Participants) | 18 | 0 | 18 | 0
  Booster Call (Phase 2) | 88.9 |  | 88.9 |

3. Primary Outcome: Percentage of Participants Who Complete Study Assessments Will be Used to Assess Feasibility and Acceptability
Description: Percentage of participants who complete study assessments, including daily surveys, one month and three month follow ups are used to assess feasibility and acceptability
Time Frame: Following intervention and follow-up assessment, measured up to 3 months
Population: Intent to treat analysis includes all participants assigned
Measure: Number; unit: percent of participants
Arm/Group | Safety Plan + Booster Text Messages + Booster Call (Group A) | Safety Plan + Booster Text Messages (Group B) | Safety Plan + Booster Call (Group C) | Safety Plan (Group D)
Number analyzed (Participants) | 18 | 22 | 18 | 22
percent of participants | 100 | 100 | 94.4 | 100

4. Primary Outcome: Satisfaction Ratings Will be Used to Assess Acceptability
Description: Satisfaction was scored by responses to two questions: How satisfied were you? on a 4 point scale, where 1 means very dissatisfied and 4 means very satisfied and how likely would you be to recommend this program to a friend in similar circumstances, on the same point scale, where 1 means definitely not and 4 means definitely yes
Time Frame: Following intervention and follow-up assessment, measured up to 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Safety Plan + Booster Text Messages + Booster Call (Group A) | Safety Plan + Booster Text Messages (Group B) | Safety Plan + Booster Call (Group C) | Safety Plan (Group D)
Number analyzed (Participants) | 17 | 22 | 16 | 22
units on a scale
  Satisfaction score | 3.59 (0.51) | 3.55 (0.51) | 3.31 (0.79) | 3.55 (0.6)
  Likelihood of recommending plan to a friend score | 3.82 (0.39) | 3.77 (0.43) | 3.38 (0.81) | 3.64 (0.49)

ADVERSE EVENTS:
Time Frame: Data on suicide attempts was collected over a 3 month period.
Description: Since all participants were hospitalized for suicide risk (ideation or attempts) to be eligible, those who were unreachable at follow-up weren't included in denominators of suicide attempt data, as they couldn't be presumed to have attempted suicide nor could they be presumed with certainty not to have attempted suicide. Thus it is most accurate to report only known data that is based on collected AEs. Non-serious Adverse Events were not collected.
Arm/Group | Safety Plan + Booster Text Messages + Booster Call (Group A) | Safety Plan + Booster Text Messages (Group B) | Safety Plan + Booster Call (Group C) | Safety Plan (Group D)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/22 | 0/18 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/15 | 2/19 | 3/14 | 3/20
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Plan + Booster Text Messages + Booster Call (Group A) (N=15) | Safety Plan + Booster Text Messages (Group B) (N=19) | Safety Plan + Booster Call (Group C) (N=14) | Safety Plan (Group D) (N=20)
Suicide Attempt (Psychiatric disorders) | 0 | 2 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT03838198/Prot_SAP_000.pdf